CLINICAL TRIAL: NCT02557243
Title: Malignant Pediatric Soft Tissue & Bone Tumors of the Extremities: A Retrospective Study
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Morsy, MD, Lecturer, Pediatric Oncology Department, Assiut University
Other Study IDs: Ped Malig Extremities; IRB00008718 (Registry Identifier: Assiut University)
Record Dates: First submitted 2015-09-21; First posted 2015-09-23 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Soft Tissue Neoplasms; Bone Neoplasms
Keywords: Childhood Cancer; Soft Tissue Tumors; Bone Tumors; Extremity Tumor; Pediatric Oncology
MeSH Terms: conditions — Soft Tissue Neoplasms; Bone Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to identify demographic & disease characteristics in pediatric oncology patients diagnosed with soft tissue & bone tumors involving the extremities & treatment outcomes in these patients.

DETAILED DESCRIPTION:
Background:

Sarcomas are a heterogeneous group of rare tumors that arise predominantly from the embryonic mesoderm. The various sarcomas include bone sarcomas (osteosarcomas and chondrosarcomas), Ewing's sarcomas, peripheral primitive neuroectodermal tumors, and soft tissue sarcomas.

Soft tissue sarcomas account for approximately 1% of adult malignancies and 7% to 15% of pediatric malignancies. Rhabdomyosarcoma is the most common soft tissue sarcoma of childhood.

There is some confusion within segments of the medical community as to the precise meaning of "soft tissue." The soft tissue of the human body includes all extraskeletal tissue that is neither epithelial, hematopoietic (marrow derived blood elements), nor parenchymal (constituent of a visceral organ). The nervous system is divided such that neither the glial nor the central neuronal elements are considered to be soft tissue, though by convention the peripheral nervous system is. In sum, the soft tissues consist of adipose tissue, fibrous tissue, musculature, vascular structures, and peripheral nerves.

About 50% to 60% of sarcomas occur in the extremities, and although they are rare, they are responsible for more deaths than testicular cancer, Hodgkin's disease, and thyroid cancer combined.

Patients & Methods:

From January 2000 till December 2015, retrieval & analysis of the medical records of pediatric patients with soft tissue & bone tumors involving the extremities will be made at the pediatric oncology department, South Egypt Cancer Institute which represents the largest referral center in Upper Egypt. These data will be categorized according to demographic characteristics, clinico-pathologic features, treatment modalities received, and outcomes of treatments in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age less than 19 years.
* Patients diagnosed with bone & soft tissue neoplasms involving the extremities.

Exclusion Criteria:

* Patients whose age more than 19 years.
* Patients diagnosed with bone & soft tissue neoplasms not involving the extremities.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric cancer patients, those diagnosed with bone & soft tissue neoplasms involving the extremities, in the period from 2000 January till 2015 December, and received treatment at the pediatric oncology department, their medical records will be retrospectively reviewed for data collection.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2016-01; Primary Completion 2019-11 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | Participants will be retrospectively followed forward in time from the date of initiation of treatment till the primary completion date of the study, an expected average of 5 years
  Time from the date of initiation of treatment until death from any cause
Event Free Survival (EFS) | Participants will be retrospectively followed forward in time from the date of initiation of treatment till the primary completion date of the study, an expected average of 5 years
  Time from the date of initiation of treatment until disease progression, or death for any reason.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Bakotic, B. W. (2001).
- [Background] Cormier JN, Pollock RE. Soft tissue sarcomas. CA Cancer J Clin. 2004 Mar-Apr;54(2):94-109. doi: 10.3322/canjclin.54.2.94. PMID 15061599
- [Background] Sondak, V. (2000).